CLINICAL TRIAL: NCT05521126
Title: The Use of Micro-Doppler Radar to Identify Service Members at Risk for Musculoskeletal Injury: A Gold Standard Comparison
Brief Title: Micro-Doppler Radar: A Gold Standard Comparison
Status: Active, not recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Lebanon Valley College (Unknown)
Responsible Party: Principal Investigator, Cayce Onks, Associate Professor of Family Medicine and Orthopaedics, Milton S. Hershey Medical Center
Other Study IDs: STUDY00020118; CDMRP-OR210069 (Other Grant/Funding Number: U.S. Army Medical Research Acquisition Activity)
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-04

CONDITIONS: Musculoskeletal Injury; Anterior Cruciate Ligament Injuries
Keywords: musculoskeletal injury; anterior cruciate ligament injury; anterior cruciate ligament repair; micro-Doppler radar; motion capture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- high risk/ACL repair cohort: The high risk cohort will be subjects who have had an ACL reconstruction procedure 9-24 months prior to enrollment.
- control group: The control group will be individuals who have not had an ACL reconstruction procedure.

SUMMARY:
The purpose of this study is to see if the study team can use micro-Doppler signal (MDS) technology to determine if someone has had an anterior cruciate ligament (ACL) reconstruction. The investigators will do this by comparing the movement data from a group of people who have had the surgery with a group who has not had the surgery to see if the micro-Doppler radar technology can accurately and predictably tell the difference.

DETAILED DESCRIPTION:
The objective of this research is to validate that radar MDS can accurately and predictably differentiate individuals at high-risk for MSKI from those who are low risk. The investigators hypothesize that MDS will identify individuals at a high-risk for MSKI more accurately than the gold-standard MC technologies. To test this hypothesis, the investigators propose a case control study that will compare adults who have undergone ACL reconstruction to a control group of healthy adults that has not. Patients who have undergone ACL reconstruction have a 6-24% chance of either re-tearing their ACL or having a subsequent knee surgery on either side within two years of successful completion of surgery and post-surgical rehabilitation. Despite being released for full activities, little is known about what makes this group at high-risk for re-tear. As such, the investigators will use this patient population as a model for identifying an at-risk population for musculoskeletal injury (MSKI). The researchers will simultaneously collect radar micro-Doppler signals and biomechanical motion capture (MC) data in a state-of-the-art human movement lab. Participants will be asked to perform a series of functional activities that will be captured by both the MDS radar and MC systems. The data sets will then be analyzed independently.

ELIGIBILITY:
Inclusion Criteria:

High risk cohort

* age 18-40
* history of ACL reconstruction
* no current musculoskeletal injuries
* ACL repair between 9 and 24 months prior to recruitment

Control cohort

* age 18-40
* never had lower extremity surgery

Exclusion Criteria:

High risk cohort

* age <18 or >40
* pregnancy
* institutionalization
* history of cerebral vascular accident
* unable to provide informed consent
* inability to perform study activities
* history of hip or knee replacement
* inability to walk or jump without a limp
* current neuromuscular disease
* any surgery in the last 6 months

Control cohort

* age < 18 or > 40
* pregnancy
* institutionalization
* history of Cerebral Vascular Accident
* unable to provide informed consent
* inability to perform study activities
* history of knee or hip replacement
* inability to walk or jump without a limp
* current neuromuscular disease
* history of lower extremity surgery
* any surgery in the last 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ACL repair cohort: Penn State Health Bone and Joint clinic
  control cohort: Penn State University/College of Medicine students and employees, Lebanon Valley College students, community sample
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
accuracy and predictability of MDS differentiation between ACL repair and control group | Day 1
  The investigators hypothesize that MDS will differentiate subjects who have recovered from an ACL reconstruction from a control cohort with accuracy and predictability. Participants will perform drop jumps, sit to stand, and walk on a treadmill in the presence of the micro-Doppler radar. MDS will be obtained for the ACL group as well as control. The micro-Doppler signature projection algorithm (mD-SPA) will then be applied to the data sets showing what percentage of the MDS are successfully classified to the ACL group versus control.

SECONDARY OUTCOMES:
accuracy of MDS differentiation between ACL repair and control groups versus the motion capture system | Day 1
  The investigators hypothesize that MDS will differentiate between the ACL group versus the control group with greater accuracy compared with the MC system. MDS will show greater sensitivity and specificity for correct classification compared with the gold standard MC. Participants will perform drop jumps, sit to stand, and walk on a treadmill while collecting simultaneously the motion capture data and MDS. The data sets will then be analyzed separately and the sensitivity and specificity of each system will be compared.
ability of micro-Doppler radar and deep learning algorithms to automatically produce predictive data | Day 1
  The investigators hypothesize that by incorporating several deep learning algorithms that can extract high-level deep features automatically through hierarchical architectures, the system will be able to automatically produce predictive data that will not require specialized knowledge to operate. This will allow the system to be used by medical assistants or medical technicians who have no expertise in interpretation of the radar MDS. The investigators will accomplish this by applying numerous deep learning algorithms to the MDS to determine which algorithms most accurately and automatically classify the ACL group from control.

CONTACTS AND LOCATIONS:
Overall Officials: Cayce A Onks, DO, MS, Principal Investigator — Milton S. Hershey Medical Center
Locations (2):
- United States (2):
  - Lebanon Valley College, Annville, Pennsylvania
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania